CLINICAL TRIAL: NCT00572533
Title: Intelligent Control Approach to Anemia Management (AIM 4)
Brief Title: Intelligent Control Approach to Anemia Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Adam Edward Gaweda, Associate Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: K25DK072085 (NIH); K25DK072085 (NIH); 1K25DK072085-01A2 (NIH)
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Results first posted 2012-12-20 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: End-Stage Renal Disease
Keywords: End-Stage Renal Disease; Chronic Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Adenosine Monophosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): ESA Dose Adjustment per standard Anemia Management Protocol
  Interventions: Other: ESA Dose Adjustment per standard Anemia Management Protocol
- Treatment (Experimental): ESA Dose Adjustment per "Smart Anemia Manager" Algorithm
  Interventions: Other: ESA Dose Adjustment per "Smart Anemia Manager" Algorithm

INTERVENTIONS:
Other: ESA Dose Adjustment per standard Anemia Management Protocol — Amount of ESA dose adjustment in Units per week guided by standard Anemia Management Protocol in use at the facility
  Other Names: AMP
  Arms: Control
Other: ESA Dose Adjustment per "Smart Anemia Manager" Algorithm — Amount of ESA dose adjustment in Units per week individualized to subject's dose-response profile guided by "Smart Anemia Manager" algorithm
  Other Names: SAM
  Arms: Treatment

SUMMARY:
First clinical evaluation of "Smart Anemia Manager" algorithm.

DETAILED DESCRIPTION:
The purpose of this single-center study is to test whether "Smart Anemia Manager" algorithm improves Hemoglobin stability compared to standard Anemia Management Protocol. Study site: Kidney Disease Program dialysis facility, University of Louisville, Louisville, KY.

ELIGIBILITY:
Inclusion criteria:

1. ages 18 to 80,
2. receiving dialysis treatment,
3. receiving or expected to receive ESA treatment,
4. adequacy of dialysis Kt/V >= 1.2,
5. adequate iron stores (Ferritin > 200 ng/mL, TSat > 20%).

Exclusion criteria:

1. life expectancy less than 12 months,
2. frequent uncontrolled blood loss,
3. frequent dialyzer clotting,
4. frequent access related problems,
5. active infections,
6. severe cardiac disability,
7. coronary bypass within three months prior to the study
8. documented resistance to ESA
9. bone marrow suppression due to HIV, leukemia, or pharmacologic agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam E Gaweda, Ph.D., Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Kidney Disease Program, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Treatment
Started | 31 | 31
Completed | 24 | 28
Not Completed | 7 | 3
Not completed — Death | 4 | 1
Not completed — Received Kidney Transplant | 2 | 1
Not completed — Social Issues | 1 | 0
Not completed — Transfer out of Facility | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Treatment | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 27 | 51
  >=65 years | 7 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (10) | 57 (9) | 57 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 22 | 20 | 42
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 21 | 41
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 62
Diabetes [Number; unit: Participants] — Number of subjects with diagnosed diabetes
  Participants
    Diabetes | 17 | 18 | 35
    No Diabetes | 14 | 13 | 27
Congestive Heart Failure (CHF) [Number; unit: Subjects] — Number of subjects with diagnosed CHF
  Subjects
    CHF | 6 | 8 | 14
    No CHF | 25 | 23 | 48
Vascular Access Type [Number; unit: Participants] — Number of patients with specific vascular access type
  Participants
    Fistula | 20 | 21 | 41
    Catheter | 6 | 3 | 9
    Graft | 5 | 7 | 12
Hemoglobin (g/dL) [Mean (Standard Deviation); unit: g/dL] — Hemoglobin concentration in March 2011
  g/dL | 11.2 (1.4) | 11.3 (1.0) | 11.3 (1.2)
ESA dose [Mean (Standard Deviation); unit: IU/week/subject] — ESA dose across group in March 2011
  IU/week/subject | 4,645 (7,468) | 5,290 (7,751) | 4,968 (7,555)

OUTCOME MEASURES:

1. Primary Outcome: Percent Hb 10-12 g/dL
Description: Percentage of Hemoglobin concentrations measured (once per month) between 10 and 12 g/dL.
Time Frame: 12 months
Population: Intent-To-Treat Analysis, Missing Data Excluded
Measure: Number; unit: Percent
Arm/Group | Control | Treatment
Number analyzed (Participants) | 31 | 31
Percent | 61.9 | 72.5

2. Secondary Outcome: Percent Hb < 10 g/dL
Description: Percentage of Hemoglobin concentrations measured (once per month) less than 10 g/dL.
Time Frame: 12 months
Population: Intent-To-Treat Analysis, Missing Data Excluded
Measure: Number; unit: Percent
Arm/Group | Control | Treatment
Number analyzed (Participants) | 31 | 31
Percent | 24.7 | 11.8

3. Post Hoc Outcome: Transfusion Events
Description: Number of Transfusion Events
Time Frame: 12 months
Population: Intent-To-Treat, Missing Data Excluded
Measure: Number; unit: Events
Arm/Group | Control | Treatment
Number analyzed (Participants) | 31 | 31
Events | 13 | 6

4. Secondary Outcome: Percent Hb > 12 g/dL
Description: Percentage of Hemoglobin concentrations measured (once per month) greater than 12 g/dL.
Time Frame: 12 months
Population: Intent-To-Treat, Missed Data Excluded
Measure: Number; unit: Percent
Arm/Group | Control | Treatment
Number analyzed (Participants) | 31 | 31
Percent | 13.4 | 15.7

5. Secondary Outcome: Mean Hb
Description: Mean Hemoglobin concentration over follow-up period
Time Frame: 12 months
Population: Intent-To-Treat Analysis, Missing Data Excluded
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Control | Treatment
Number analyzed (Participants) | 31 | 31
g/dL | 10.7 (1.5) | 11.0 (1.2)

6. Secondary Outcome: ESA Dose
Description: Mean ESA dose per patient-week. ESA used: Epoetin Alfa (IV)
Time Frame: 12 months
Population: Intent-to-Treat Analysis, Missing Data Excluded
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Control | Treatment
Number analyzed (Participants) | 31 | 31
IU | 3,033 (3,592) | 3,704 (5,221)

7. Post Hoc Outcome: Subjects Receiving Transfusion
Description: Number of Subjects receiving Transfusion
Time Frame: 12 months
Population: Intent-To-Treat, Missing Data Excluded
Measure: Number; unit: Participants
Arm/Group | Control | Treatment
Number analyzed (Participants) | 31 | 31
Participants | 8 | 5

8. Post Hoc Outcome: RBC Units Transfused
Description: Total number of RBC units transfused
Time Frame: 12 months
Population: Intent-To-Treat, Missing Data Excluded
Measure: Number; unit: RBC Units
Arm/Group | Control | Treatment
Number analyzed (Participants) | 31 | 31
RBC Units | 31 | 21

ADVERSE EVENTS:
Time Frame: 04/01/2011 - 03/31/2012
Arm/Group | Control | Treatment
Serious Adverse Events (participants affected / at risk) | 19/31 | 18/31
Other Adverse Events (participants affected / at risk) | 17/31 | 16/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=31) | Treatment (N=31)
Composite Safety Event (ACM, MI, CVA, CHF) (General disorders) | 6 (10) | 10 (11) — All-Cause Mortality, Myocardial Infarction, Cerebrovascular Accident, Congestive Heart Failure
Hospitalization (General disorders) | 18 (39) | 18 (41) — All-Cause Hospitalization (includes hospitalization due to Composite Safety Event)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=31) | Treatment (N=31)
Vascular Access Event (Surgical and medical procedures) | 17 (27) | 16 (38)
Infection (General disorders) | 5 (8) | 6 (10)

LIMITATIONS AND CAVEATS:
1. Single-center design
2. Small sample size
3. Homogenous population
4. Only maintenance dosing phase tested

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No